CLINICAL TRIAL: NCT05250856
Title: A Phase 1b/2a Study to Evaluate the Safety, Tolerability, and Pharmacodynamics of CNP-201 in Subjects Ages 16-55 With Peanut Allergy
Brief Title: CNP-201 in Subjects With Peanut Allergy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lagging Enrollment and Administrative Reasons
Sponsor: COUR Pharmaceutical Development Company, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CNP-201-5.002
Record Dates: First submitted 2022-02-11; First posted 2022-02-22 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Peanut Allergy
Keywords: Allergy; Food Allergy
MeSH Terms: conditions — Peanut Hypersensitivity; Hypersensitivity; Food Hypersensitivity

STUDY DESIGN:
Intervention Model Description: The study was designed with multiple ascending doses of CNP-201 in a Dose Escalation Phase, with the goal of identifying a safe and tolerable dose level to be evaluated further in a larger number of subjects in a Dose Expansion Phase. However, the study was terminated for administrative reasons and lagging enrollment within the Dose Escalation Phase.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- CNP-201 1 mg (Experimental): intravenous infusion on Day 1 and Day 8: 1 mg CNP-201
  Interventions: Drug: CNP-201
- CNP-201 2 mg (Experimental): intravenous infusion on Day 1 and Day 8: 2 mg CNP-201
  Interventions: Drug: CNP-201
- CNP-201 4 mg (Experimental): intravenous infusion on Day 1 and Day 8: 4 mg CNP-201
  Interventions: Drug: CNP-201
- CNP-201 8 mg (Experimental): intravenous infusion on Day 1 and Day 8: 8 mg CNP-201
  Interventions: Drug: CNP-201
- Placebo (Placebo Comparator): 200 ml intravenous infusion on Day 1 and Day 8: CNP-201 Placebo
  Interventions: Drug: CNP-201; Drug: Placebo

INTERVENTIONS:
Drug: CNP-201 — CNP-201 is comprised of purified peanut extract (PPE) drug substance dispersed within a negatively charged polymer matrix of poly (lactic-co-glycolic acid) (PLGA) particles at a target concentration of ~5 μg of PPE per mg of PLGA.
Drug: Placebo — Placebo, (0.9% Sodium Chloride for IV infusion)
  Arms: Placebo

SUMMARY:
This study is a Phase 1b/2a clinical trial to assess the safety, tolerability, and pharmacodynamics of multiple ascending doses (Escalation Phase) of CNP-201 with the goal of identifying a safe and tolerable dose level to be evaluated further in a larger number of subjects (Expansion Phase).

DETAILED DESCRIPTION:
The Escalation Phase will consist of multiple cohorts (4 subjects per cohort) to identify a safe and tolerable dose(s). The Expansion Phase will consist of up to 40 additional subjects who will receive either a Placebo or CNP-201 at a safe and tolerable dose as determined from the Escalation Phase. One or more dose levels may be explored in the Expansion Phase.

Subjects who meet all inclusion and no exclusion criteria at screening will be enrolled into the study.

In the Escalation Phase, each cohort of four (4) subjects will receive CNP-201 by intravenous (IV) infusion on Days #1 and #8. Subjects in the Expansion Phase will be randomized in a 1:1 ratio to receive either a safe and tolerable dose level of CNP-201 identified in the Escalation Phase or Placebo (0.9% Sodium Chloride for injection).

Subjects will remain in the clinic on Days #1 and #8 from the time of admission (prior to administration of CNP-201 or Placebo) through the final procedure conducted 4-hours post-dose that same day unless an infusion reaction, anaphylaxis, or other adverse event requires an extended duration of monitoring. Subjects will be discharged if safety parameters are acceptable to the investigator. Seven (7) days after the second administration of CNP-201 or Placebo, subjects must return to the clinic for collection of safety labs, PD measurements, and assessment of AEs and medication changes.

Subjects will continue to be followed for safety, and tolerability during a 52-day Post-Dosing period.

On Day 60, subjects will return to the clinic for collection of immune safety labs, PD measurements and to undergo Day 1 a Double-Blind, Placebo-Controlled Food Challenge (DBPCFC) consisting of peanut and placebo (oat) challenges. On Day 61, subjects will return to the clinic to undergo Day 2 of the DBPCFC and final assessment of AEs and medication changes.

The total duration of the study for an individual subject is approximately 67 days: 7 days for Screening; 8 days for CNP-201 or Placebo dosing; and 52 days post-dosing evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Men and non-pregnant women, ages 16 to 55 years inclusive.
2. Subjects with physician-diagnosed peanut allergy or documented history of peanut allergy. Note: If subject does not have documented history in their medical record but is reasonably suspected of having peanut allergy and is deemed to otherwise be a good candidate for this trial, the screen testing (peanut specific IgE, SPT, etc.) may be used to establish the peanut allergy and the PI may subsequently document the peanut allergy to fulfill this inclusion criterion.
3. Subjects with weight ≥ 31.25 kg at Screening. Subjects who fall outside of this range may be included at the discretion of the investigator.
4. Subjects with a documented history of non-severe anaphylaxis (Grade ≤ 3) to peanuts, including mild wheezing or dyspnea without hypoxia.
5. Subjects with peanut specific IgE > 5 kU/L as measured by ImmunoCAP at Screening. Subjects who have previously been on OIT for peanut allergy and who do not have peanut specific IgE ≥ 5 kU/L as measured by ImmunoCAP at Screening may be included at the discretion of the investigator, OR Subjects with a positive skin prick test (SPT) to peanut with a change in wheal diameter ≥ 3 mm as compared to a negative control (50% glycerin) at Screening. Subjects who have previously been on OIT for peanut allergy and who do not have a positive skin prick test (SPT) to peanut with a change in wheal diameter ≥ 3 mm at Screening may be included at the discretion of the investigator.
6. Subjects who are self-reported to be on a peanut free diet with no suspected peanut exposure, including any peanut food challenge, for at least 14 days prior to Screening and agreement to continue restriction to peanut exposure during the study.
7. Female subjects and male subjects and their female spouse/partners who are willing to practice a highly effective method of contraception that may include, but is not limited to, abstinence, sex only with persons of the same sex, monogamous relationship with vasectomized partner, vasectomy, hysterectomy, bilateral tubal ligation, licensed hormonal methods, intrauterine device (IUD), or use of spermicide combined with a barrier method (e.g., condom, diaphragm) starting at Screening and continuing to Day 60.
8. Female subjects who agree to not breastfeed starting at initial Screening and continuing to Day 60.
9. Female subjects who agree to not donate ova starting at initial Screening and continuing to Day 60.
10. Subjects who are willing and able to provide Institutional Review Board (IRB) approved written informed consent.
11. Subjects who are willing to perform and comply with all study procedures.
12. Male subjects who agree to not donate sperm starting at Screening and continuing to Day 60.

Exclusion Criteria:

1. Subjects with history of severe anaphylaxis to peanuts defined as neurological compromise or requiring intubation.
2. Subjects with peanut specific IgE ≥ 100 kU/L as measured by ImmunoCAP at Screening.
3. Subjects who have received administration of vaccinations in the following timeframe:

   * Any live vaccine (other than intranasal Influenza) within 28 days prior to Screening.
   * Any subunit vaccine within 14 days prior to Screening.
4. Any COVID-19 vaccine within 14 days prior to Screening. Subjects who have received the first dose of any COVID-19 vaccine may not screen for the study until 14 days following their last dose of the vaccine if applicable.
5. Any planned vaccination prior to Day 15.
6. Subjects in build-up phase of immunotherapy for aeroallergens or venom. Individuals tolerating maintenance aeroallergen or venom immunotherapy at Screening can be enrolled.
7. Subjects with relative contraindication or inability to use epinephrine auto-injector.
8. Subjects who have used the following drug(s) within 2 months prior to Screening: Th2 cytokine inhibitors, thromboxane A2 synthesis inhibitors, thromboxane A2 receptor antagonists, β-blockers, angiotensin-converting enzyme inhibitors, and/or angiotensin-receptor blockers unless, in the investigator's opinion, the underlying condition being treated by the drug is well controlled and the drug dose and frequency is not expected to interfere with the mechanism of action of CNP-201 as determined in consultation with the sponsor.
9. Subjects who have used biologics and/or immune modulators (including but not limited to anti-TNFα antibody and anti-IgE monoclonal antibody) within three months prior to Screening.
10. Subjects with a history of allergic reactions such as anaphylactic shock, angioedema with airway constriction, or hypotension caused by food other than peanut and/or medical products.
11. Subjects with positive test results for hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or human immunodeficiency virus (HIV) antigen/ antibody as determined at Screening.
12. Subjects who are immunocompromised, including those receiving immunosuppressive doses of corticosteroids (more than 20 mg of prednisone given daily or on alternate days for 2 weeks or more within 6 months prior to Screening, any dose of corticosteroids within 30 days of Screening, or high dose inhaled corticosteroids [> 960 μg/day of beclomethasone dipropionate or equivalent]) or other immunosuppressive agents.
13. Subjects with a history of unstable angina pectoris, cardiac disease or dysrhythmias, severe chronic lung disease, or any other chronic medical condition that which in the opinion of the investigator, would pose a significant health threat in the event of anaphylaxis/treatment of anaphylaxis.
14. Subjects with active eosinophilic esophagitis (EoE) or other eosinophilic gastrointestinal disease.
15. Subjects with clinically significant abnormality on electrocardiogram (ECG) at Screening that, in the investigator's opinion, makes the subject unsuitable for study participation.
16. Subjects with active malignancy, or history of malignancy or chemotherapy within the past 5 years other than history of localized or surgical removal of focal skin cancer, or cervical cancer in situ treated successfully in the past by local treatment (including but not limited to cryotherapy or laser therapy) or by hysterectomy.
17. Subjects with a mental condition such as schizophrenia, bipolar disorder, major depressive disorder, generalized anxiety disorder, panic disorder/attacks, or subjects who have received drug(s) for the treatment of dementia.
18. Subjects with severe or poorly controlled (resistant to appropriate medical intervention) atopic disease including atopic dermatitis, generalized eczema, allergic rhinitis and/or urticaria.
19. Subjects with tryptase values outside of the normal reference range.
20. Subjects with severe or uncontrolled/difficult to control asthma/wheezing, defined by at least one of the following criteria:

    * Global Initiative for Asthma (GINA) 2020: Personalized management to control symptoms and minimize future risk requiring treatment Steps 4 or 5 (Appendix 3) OR;
    * Forced expiratory volume in 1 second (FEV1) < 80% of predicted, or ratio of FEV1 to forced vital capacity (FEV1/FVC) < 75% of predicted, with or without controller medications (only those able to reliable perform spirometry. If unable to do spirometry, PEF of > 80% is acceptable OR;
    * One overnight admission to a hospital in the past year for asthma OR;
    * Emergency room visit for asthma within 6 months prior to Screening OR;
    * History of two or more systemic corticosteroid courses within 6 months of Screening or one course of systemic corticosteroids within 3 months of Screening to treat asthma/wheezing OR;
    * Prior intubation/mechanical ventilation for asthma/wheezing.
21. Subjects who have received an investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to Screening.
22. Subjects with any condition which, in the investigator's opinion, makes the subject unsuitable for study participation: Past or current medical problems, history of other chronic diseases requiring therapy, findings from physical assessment, or abnormalities in clinical laboratory testing that are not listed above, which in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements, or that may impact the quality or interpretation of the data obtained from the study.
23. Subjects with a known sensitivity to any components of CNP-201 (PLGA, sucrose, mannitol, or sodium citrate).

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 15 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Frequency of Adverse Events (AEs) and Serious Adverse Events (SAEs) | through Study Completion, an average of 67 Days
  Frequency tables will be presented by treatment group for all AEs and SAEs by System Organ Class (SOC) and Preferred Term (PT). Frequency tables will also be produced by treatment group for AEs leading to discontinuation from TP and study, by severity, and by causality. No formal statistical testing will be done.
Serum Cytokines (TNF-α, IL-2, IL-6, IL-8, IL-1β, MCP-1, MIP-1β, MIP-1α, IFN-γ, and IL-12p70) | Baseline (Day 1 pre-dose) through Day 60, an average of 52 Days
  Summary statistics will be presented for the change from baseline values for Serum Cytokines (TNF-α, IL-2, IL-6, IL-8, IL-1β, MCP-1, MIP-1β, MIP-1α, IFN-γ, and IL-12p70)

SECONDARY OUTCOMES:
Change in the ratio of peanut specific IgE to IgG | Baseline (Day 1 pre-dose) through Day 60, an average of 52 Days
  The mean change in the ratio of peanut specific IgE to IgG as measured by ImmunoCap assay from Baseline (Screening) to Visit 5 within CNP-201 and Placebo treatment groups will be analyzed
Change in peanut specific IgE between CNP-201 and Placebo | Baseline (Day 1 pre-dose) through Day 60, an average of 52 Days
  The mean change of peanut specific IgE to IgG as measured by ImmunoCap assay from Baseline (Screening) to Visit 5 within CNP-201 and Placebo treatment groups will be analyzed
Difference in percentage of subjects who pass a DBPCFC | At Day 60
  Difference in percentage of subjects who pass a DBPCFC (do not reach an eliciting dose at or before the 2000 mg dose level, 4043 mg cumulative) between placebo and CNP-201 at Day 60 and at Day 180
Change in the proportion of peanut specific Th2a+ T cells | Baseline (Day 1 pre-dose) through Day 15, an average of 15 Days
  Change in the proportion of peanut specific Th2a+ T cells (peanut specific Th2a+ cells / total peanut specific T cells) following ex vivo stimulation of PBMCs between placebo and CNP-201 at baseline and at Day 15
Change in the effective concentration at 50% of maximal basophil activation (EC50) | Baseline (Day 1 pre-dose), at Day 15, and at Day 60
  Change in the effective concentration at 50% of maximal basophil activation (EC50) as measured by a Basophil Activation Test (CD203c+/CD63+/- basophil activation) between placebo and CNP-201 at baseline and at Day 60 and at Day 180
Change in the proportion of peanut specific T regulatory cells (peanut specific T regulatory cells / peanut specific CD4+ effector memory cells) | Baseline (Day 1 pre-dose) and at Day 15
  Change in the proportion of peanut specific T regulatory cells (peanut specific T regulatory cells / peanut specific CD4+ effector memory cells) following ex vivo stimulation of PBMCs between placebo and CNP 201 at baseline and at Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Jerry Staser, Study Director — COUR Pharmaceuticals
Locations (17):
- United States (17):
  - AllerVie Clinical Research, Birmingham, Alabama
  - Long Beach Clinical Trials, LLC, Long Beach, California
  - Southern California Research, Mission Viejo, California
  - Allergy & Asthma Medicaal Group and Research Center, San Diego, California
  - Rush University Medical Center, Chicago, Illinois
  - Sneeze, Wheeze and Itch Associates, LLC, Normal, Illinois
  - Meridian Clinical Research. LLC, Overland Park, Kansas
  - Institute for Asthma & Allergy, Chevy Chase, Maryland
  - Aventiv Research, Inc, Columbus, Ohio
  - Vital Prospects Clinica Research Institute, Tulsa, Oklahoma
  - National Allergy and Asthma Research, LLC, North Charleston, South Carolina
  - Allergy Partners of North Texas Research, Dallas, Texas
  - Pharmaceutical Research & Consulting, Inc, Dallas, Texas
  - Western Sky Medical Research, El Paso, Texas
  - Tranquil Clinical and Research Consulting Services, Houston, Texas
  - Clinical Research Partners, Richmond, Virginia
  - Seattle Allergy & Asthma Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No